CLINICAL TRIAL: NCT05242601
Title: Investigation of Quality of Life in Adolescent Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Mehmet Hanifi Kaya, lecturer, Kirsehir Ahi Evran Universitesi
Other Study IDs: 27.04.2021-10775
Record Dates: First submitted 2022-01-27; First posted 2022-02-16 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — no intervention

SUMMARY:
the aim of our study is to identify independent predictors of quality of life in AIS.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is the lateral and horizontal deformity of the columna vertebralis which occurs idiopathically in adolescence ages. The aim of this study is to identify independent predictors of quality of life in AIS

ELIGIBILITY:
Inclusion Criteria:

* volunteered for the study participants were diagnosed with adolescent idiopathic scoliosis,
* between ages 10-18
* Cobb angle between 10-30 degrees
* Lenke curve type 1

Exclusion Criteria:

* non-idiopathic scoliosis,
* who had exercise contraindications
* who had previous spinal surgery
* who had orthotic treatment for scoliosis before
* who had exercise contraindications
* who had another neuromuscular
* who had cardiopulmonary and rheumateulogical problem

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: volunteered for the study participants were diagnosed with adolescent idiopathic scoliosis,
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-09-12 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Investigation of Quality of Life in Adolescent Idiopathic Scoliosis | 4 week
  Quality of life Scoliosis Research Society-22 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

REFERENCES:
- [Derived] Kaya MH, Erbahceci F, Alkan H, Kocaman H, Buyukturan B, Canli M, Buyukturan O. Factors influencing of quality of life in adolescent idiopathic scoliosis. Musculoskelet Sci Pract. 2022 Dec;62:102628. doi: 10.1016/j.msksp.2022.102628. Epub 2022 Jul 19. PMID 35872563